CLINICAL TRIAL: NCT05315440
Title: The Effectiveness of Graston Tecnique Compared to Traditional Physiotherapy to Improve Shoulder Range of Motion After Arthroscopic Cuff Repair.
Brief Title: The Effectiveness of Graston Tecnique Compared to Traditional Physiotherapy to Improve Range of Motion After Arthroscopic Cuff Repair.
Acronym: GRA-RCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0002771
Record Dates: First submitted 2021-09-14; First posted 2022-04-07 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Cuff Tear Arthropathy
Keywords: shoulder rehabilitation; range of motion; rotator cuff repair; instrument assisted soft tissue mobilitation
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: outcome assessor doesn't know allocation concealment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): The treatment of control group will be organized according to the classic protocol currently in use in our Institute which consists of:
  30 minutes of passive and active assisted mobilization guided by the therapist, 30 min of Continous passive movement in flexion and abduction and 30 minutes of electrostimulation.
  Interventions: Other: Conventional rehabilitation
- experimental group (Experimental): 30 minutes of passive and active assisted mobilization guided by the therapist associated with instrument assisted soft tissue mobilization, 30 min of Continous passive movement in flexion and abduction and 30 minutes of electrostimulation.
  Interventions: Other: graston tecnique

INTERVENTIONS:
Other: graston tecnique — Graston technique involves the use of steel tools that are used non-invasively on the skin to identify and treat areas that have stiffness or inflammation. These areas can be located with greater precision than the manual technique precisely because the instruments do not compress in contact with the patient's skin, as is the case with the physiotherapist's fingertips. Thanks to the instruments it is therefore possible to detect the areas of altered consistency and to treat them by pressing a minimum pressure.
  Other Names: instrument soft tissue mobilization
  Arms: experimental group
Other: Conventional rehabilitation — 30 minutes of passive and active assisted mobilization guided by the therapist, 30 min of Continous passive movement in flexion and abduction and 30 minutes of electrostimulation.
  Arms: control group

SUMMARY:
In shoulder rehabilitation after arthroscopic cuff repair, one of first objectives coincides with improving the range of passive movement: this process often requires considerable time of both patients and physiotherapists. This study aims to verify whether it is useful to add instruments assisted soft-tissue mobilization according to Graston Tecnique to the classic rehabilitation protocol in order to accelerate recovery times of passive range of motion.

DETAILED DESCRIPTION:
There is conflicting evidence about early versus delayed postoperative rehabilitation after arthroscopic cuff repair: early protocol seems to reduce the risk of stiffness but could increase the risk of rupture of the tendon in long time, especially for large tears; delayed protocol impose a period of shoulder immobilization (from 2 weeks to 40-day) that can promote tendons healing but could determine shoulder stiffness. Our research question is if after the delayed protocol used in our institute (40 -day immobilization period) it migh be useful to add soft-tissue mobilization assisted by instruments according to Graston Tecnique to the classic rehabilitation protocol of the shoulder in order to speed up recovery times of the passive movement range.

ELIGIBILITY:
Inclusion Criteria:

* arthroscopic rotator cuff repair
* partial lesion due to tendon degeneration (1 or 2 anchors reparation)

Exclusion Criteria:

* traumatic tendon lesions
* associated conditions as arthritis, loss of superficial sensitivity, loss of muscle tone, mental impairment, oncological conditions
* shoulder stiffness before surgery due to calcific tendonitis, adhesive capsulitis

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Passive Range of Motion Recovery of the Shoulder | after 2 weeks of treatment
  Passive Range of Motion Recovery of the Shoulder in elevation and abduction measured by digital inclinometer

SECONDARY OUTCOMES:
Reduction of pain measured by Visual Analogue Scale (VAS) | after 2 weeks of treatment
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between 0 ("no pain") and 10 ("worst pain").
Shoulder function improvement measured by Constant Murley and Dash scales | after 2 weeks of treatment
  The Constant-Murley score is a 100-points scale composed of a number of individual parameters that define the level of pain and the ability to carry out the normal daily activities of the patient. The test is divided into 4 subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion (40 points). The higher the score, the higher the quality of the function. Since the test is carried out in an acute post-surgery phase, it is not possible to carry out the evaluation of strength, which is assigned a score of zero for all patients. The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. This questionnaire is a self-report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale.The score ranges from 0 (no disability) to 100 (most severe disability).

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided